CLINICAL TRIAL: NCT07284511
Title: Fully Closed-Loop Glucose Control in Adults With Type 1 Diabetes Using Tirzepatide: a Randomized, Multi-center, Open-label, Non-inferiority, Parallel Trial
Brief Title: A Clinical Trial Using Tirzepatide to Help Adults With Type 1 Diabetes Automatically Control Their Blood Sugar
Acronym: TZP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Melissa-Rosina Pasqua (Other)
Collaborators: Breakthrough T1D (Other); Institut de Recherches Cliniques de Montreal (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Melissa-Rosina Pasqua, Principal Clinical Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026-12143
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus; T1D; T1DM; T1DM - Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Overweight or obesity in type 1 diabetes; Automated insulin delivery; Insulin pump; Continuous glucose monitoring; Tirzepatide; Mounjaro; GIP/GLP-1 receptor agonist; Dual incretin therapy; Adjunctive tirzepatide therapy; Tandem Control-IQ; Hybrid closed-loop system; Closed-loop insulin delivery; Dexcom G7
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, parallel-group clinical trial conducted at multiple centers. After a standardized run-in with the Tandem Control-IQ insulin pump and Dexcom G7 glucose sensor, adults with type 1 diabetes are randomized in balanced blocks to either adjunct tirzepatide or control. Randomization is stratified by site and baseline insulin therapy. Participants in both groups use the same automated insulin delivery system for 32 weeks. The tirzepatide group undergoes dose escalation, maintenance, and finally a no-meal-announcement phase, while the control group continues carbohydrate counting throughout. The primary analysis compares daytime (06:00-24:00) time-in-range (3.9-10.0 mmol/L) during the last four weeks using a non-inferiority framework. This design allows rigorous evaluation of whether tirzepatide enables safe omission of meal announcements while maintaining glucose control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tirzepatide group (Experimental): Participants randomized to this arm receive once-weekly subcutaneous tirzepatide in addition to use of the Tandem Control-IQ insulin pump and Dexcom G7 continuous glucose monitor. Tirzepatide is initiated at 2.5 mg weekly and increased by 2.5 mg every 4 weeks to a target dose of 10 mg weekly or the maximally tolerated dose. Dose escalation may be delayed or reduced if participants experience intolerable gastrointestinal symptoms. During Weeks 1-26, participants continue standard carbohydrate counting for all meals. Beginning in Week 27, participants stop entering carbohydrate amounts into the pump (no meal announcements) for six weeks while continuing tirzepatide at their maintenance dose. Throughout the intervention, participants undergo regular safety assessments, remote glucose data reviews, insulin-pump parameter adjustments as needed, and scheduled in-person visits to monitor metabolic, cardiovascular, and patient-reported outcomes.
  Interventions: Drug: Tirzepatide; Device: Tandem Control-IQ Automated Insulin Delivery System (with Dexcom G7 CGM); Behavioral: Carbohydrate Counting; Behavioral: No Meal Announcement
- Control group (Active Comparator): Participants randomized to the control arm use the Tandem Control-IQ automated insulin delivery system with the Dexcom G7 continuous glucose monitor, following standard-of-care diabetes management. They continue carbohydrate counting for all meals throughout the 32-week study and deliver prandial insulin boluses based on estimated carbohydrate intake, as is typical for users of hybrid closed-loop systems. No tirzepatide injections are administered. Participants receive the same device training, follow-up schedule, safety monitoring, glucose data reviews, and pump parameter adjustments as the tirzepatide arm. This arm serves as an active comparator, representing current standard therapy for type 1 diabetes with automated insulin delivery and meal announcements.
  Interventions: Device: Tandem Control-IQ Automated Insulin Delivery System (with Dexcom G7 CGM); Behavioral: Carbohydrate Counting

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide, administered as a once-weekly subcutaneous injection, initiated at 2.5 mg and escalated in 2.5-mg increments every 4 weeks to a target of 10 mg or the maximally tolerated dose, used as an adjunct therapy in adults with type 1 diabetes using the Tandem Control-IQ automated insulin delivery system.
  Other Names: Mounjaro
  Arms: Tirzepatide group
Device: Tandem Control-IQ Automated Insulin Delivery System (with Dexcom G7 CGM) — This intervention uses the Tandem t:slim X2 insulin pump with the Control-IQ automated insulin delivery algorithm, integrated with the Dexcom G7 continuous glucose monitor. The system adjusts basal insulin and delivers automated correction boluses based on real-time glucose values. All participants receive standardized training and use this system for the full 32-week study. Rapid-acting insulin compatible with Control-IQ is required. This intervention is distinguished by its use under two different operational strategies: standard carbohydrate counting in the control arm and complete omission of meal announcements during the final 6 weeks in the tirzepatide arm.
  Other Names: Control-IQ; Dexcom G7
Behavioral: Carbohydrate Counting — Participants enter the estimated carbohydrate amount for every meal and snack into the Tandem Control-IQ insulin pump to calculate and deliver prandial insulin boluses. This reflects standard use of hybrid closed-loop systems. The procedure is maintained for the entire 32-week study in the control arm and during Weeks 1-26 in the tirzepatide arm.
  Other Names: Meal Announcement
Behavioral: No Meal Announcement — Participants do not enter carbohydrate amounts or announce meals to the Tandem Control-IQ system. The pump operates without user-initiated prandial boluses, relying solely on automated basal adjustments and automated correction boluses. This intervention is implemented only in the tirzepatide arm during Weeks 27-32.
  Other Names: Omission of Carbohydrate Counting
  Arms: Tirzepatide group

SUMMARY:
This research study is testing whether a weekly medication called tirzepatide can help adults with type 1 diabetes use their insulin pump more easily, specifically by reducing or eliminating the need to count carbohydrates at meals.

People with type 1 diabetes must take insulin for life, and even with advanced insulin pumps and continuous glucose monitors, many still struggle to keep blood sugar within the target range. One of the biggest challenges is carbohydrate counting, which requires estimating the amount of carbohydrates in every meal to give the correct insulin dose.

Tirzepatide is a medication currently approved for type 2 diabetes and weight management. Early research suggests it may also help people with type 1 diabetes by lowering appetite, slowing digestion, reducing insulin needs, and smoothing after-meal blood sugar rises.

This study will include 105 adults with type 1 diabetes at centers in Canada and Switzerland. Everyone will use the Tandem Control-IQ insulin pump with a Dexcom G7 continuous glucose monitor. Participants are randomly assigned to one of two groups:

Tirzepatide group:

Participants receive weekly tirzepatide injections. After the dose is gradually increased over 12 weeks, they will eventually try using their insulin pump without entering carbohydrate amounts at meals.

Control group:

Participants continue their usual therapy and keep counting carbohydrates for their mealtime insulin doses.

The main goal of the study is to learn whether people taking tirzepatide can safely maintain good blood sugar control without counting carbs, compared with standard care. All participants will attend several clinic visits and share their glucose, insulin, and health data throughout the 32-week trial. Some centers will also conduct heart/fitness, or body-composition tests.

As with any medication, tirzepatide may cause side effects such as nausea, vomiting, diarrhea, or decreased appetite. Rare but serious risks like gallbladder disease or pancreatitis are also monitored. Pregnancy must be avoided during the trial.

Overall, this study aims to understand whether adding tirzepatide to automated insulin delivery can simplify diabetes management, reduce burden, and maintain safe and effective glucose control for adults living with type 1 diabetes.

DETAILED DESCRIPTION:
Current diabetes technology, including hybrid automated insulin delivery systems like the Tandem Control-IQ paired with the Dexcom G7 continuous glucose monitor, improves glucose control but still relies heavily on patients entering carbohydrate amounts before eating, a task that is difficult, error-prone, and often stressful.

Tirzepatide, which is approved for type 2 diabetes and weight management, works by slowing digestion, lowering appetite, reducing insulin requirements, and improving after-meal glucose spikes, and early evidence suggests it may offer similar benefits in type 1 diabetes. This study is designed to determine whether adding once-weekly tirzepatide injections to a commercially available automated insulin delivery system can make diabetes management easier for adults with type 1, particularly by reducing or eliminating the need to count carbohydrates at meals.

In this 32-week trial, 105 adults will be randomly assigned to receive tirzepatide or no tirzepatide while all participants use the Control-IQ system. Those receiving tirzepatide will gradually increase their dose over 12 weeks, continue counting carbohydrates until week 26, and then stop announcing meals entirely for the final 6 weeks, while the control group will count carbohydrates throughout.

Across the study, participants will attend scheduled clinic visits, complete remote follow-ups, undergo laboratory tests, and, depending on the site, may complete heart function tests, body-composition scans, fitness testing, or gastric emptying assessments. Researchers will compare glucose control, insulin needs, weight, metabolic markers, meal patterns, and patient-reported outcomes between groups, with the primary goal of determining whether glucose management without carbohydrate counting is not worse than (non-inferior to) standard carbohydrate counting.

The study also closely monitors safety, as tirzepatide can cause nausea, vomiting, diarrhea, decreased appetite, and rare complications such as gallbladder disease or pancreatitis. Overall, this research aims to learn whether combining tirzepatide with automated insulin delivery can safely simplify diabetes management, reduce treatment burden, and improve metabolic outcomes for adults living with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of type 1 diabetes for ≥ 1 year, per investigator judgment (confirmatory C-peptide and autoantibodies not required).
* A BMI ≥ 27 kg/m2.
* HbA1c > 6.5%, and < 12%.
* Current therapy: multiple daily injections or insulin pump.
* Willingness to use Tandem Control IQ insulin pump system with the use of rapid or ultra rapid-acting insulins compatible with Tandem Control-IQ pump (e.g. Fiasp is not compatible)
* Active carbohydrate counting for prandial insulin dosing.
* Individuals of childbearing potential must be using or agree to use an effective birth-control method. Childbearing potential refers to participants of the female sex post-menarche who have not reached menopause and who do not have a medical condition causing sterility (e.g., hysterectomy). Post-menopausal state refers to the absence of menses for 12 months without any alternative cause.

Exclusion Criteria:

* Use of GLP1-RAs within the last four weeks.
* Use of antihyperglycemic agents other than insulin or metformin within the last 2 weeks.
* Planned or ongoing pregnancy.
* Breastfeeding.
* Severe hypoglycemia requiring hospitalization in the past 2 months. Severe hypoglycemia is defined as requiring the assistance of another person, due to altered consciousness, to administer carbohydrates, glucagon, or other resuscitative actions.
* Diabetic ketoacidosis within the last 2 months.
* History of acute or chronic pancreatitis.
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2.
* Severe renal impairment with eGFR <30 mL/min/1.73 m2 (CKD-EPI), measured within the last four months.
* Clinically significant proliferative diabetic retinopathy or gastroparesis, as per the judgment of the investigator.
* Current or ≤ 1 month use of supraphysiological doses of oral or intravenous glucocorticoids.
* History of bariatric surgery within the last 6 months.
* Medical or psychiatric illness likely to interfere with participation (e.g. cirrhosis, active cancer, decompensated schizophrenia), per investigator judgment.
* Inability or unwillingness to comply with safe diabetes management practices, in the view of the investigator.
* Any safety concern that, in the investigator's judgment, precludes participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Daytime Time-in-Range | During the final 6 weeks of the study
  The primary outcome is the percentage of daytime hours (06:00-24:00) during which participants' glucose levels, measured by the Dexcom G7 continuous glucose monitor, fall within the target range of 3.9-10.0 mmol/L.

SECONDARY OUTCOMES:
Weight | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study
  Change in body weight to assess the effects of tirzepatide on body composition. Weight is measured in kilograms.
Height | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study.
  Change in height to assess the effects of tirzepatide on body composition. Height is measured in meters.
Body Mass Index | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study
  Change in BMI to assess the effects of tirzepatide on body composition. BMI is measured in kilograms per square meter.
Waist circumference | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study
  Change in waist circumference to assess the effects of tirzepatide on body composition. Waist circumference is measured in centimetres.
Waist-to-Hip Ratio | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study.
  Change in waist-to-hip ratio to assess the effects of tirzepatide on body composition. Waist-to-Hip Ratio is measured by dividing the waist circumference by the hip circumference. It is unitless.
Systolic Blood Pressure | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study.
  Change in systolic blood pressure to evaluate the cardiovascular effects of tirzepatide. Systolic blood pressure is measured in millimetres of mercury.
Diastolic Blood Pressure | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study.
  Change in diastolic blood pressure to evaluate the cardiovascular effects of tirzepatide. Diastolic blood pressure is measured in millimetres of mercury.
Resting Heart Rate | At enrollment, Week 8, Week 16, Week 24, and Week 32, At Week 8 and Week 16 post-study.
  Change in resting heart rate to assess the cardiovascular effects of tirzepatide. Resting heart rate is measured in beats per minute.
Insulin-related measures | Continuously from randomization through Week 32, with primary analysis focused on Weeks 27-32, At Week 8 and Week 16 post-study.
  Daily insulin requirements, including basal insulin, bolus insulin, and total insulin units per day, recorded through the insulin pump.
  Total insulin use normalized to body weight (units/kg/day) to assess treatment-related changes in insulin sensitivity.
  Carbohydrate amounts entered for bolus dosing (control arm and Weeks 1-26 of tirzepatide arm).
Glucose outcomes | Continuously collected from randomization through Week 32, with key comparisons during Weeks 23-26 and Weeks 27-32, At Week 8 and Week 16 post-study.
  Percentage of CGM readings within 3.9-10.0 mmol/L, 3.9-7.8 mmol/L, <3.9 mmol/L, <3.0 mmol/L, >10.0 mmol/L, and >13.9 mmol/L, as well as mean glucose, glucose standard deviation, and glucose coefficient of variation.
Glycated Hemoglobin (HbA1c) | At enrollment, mid-study at Week 16, and at the end-of-study visit at Week 32, At Week 8 and Week 16 post-study.
  Change in glycated hemoglobin (HbA1c) to assess overall glycemic control over the study period.
Estimated Glomerular Filtration Rate | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in estimated glomerular filtration rate. eGFR is measured in millilitres/minute/body surface.
Serum Creatinine | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in serum creatinine. Serum creatinine is measured in umol/L.
Albumin-to-Creatinine Ratio | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in urinary albumin-to-creatinine ratio. Urinary albumin-to-creatinine ratio is measured in mg/mmol.
Lipid Panel (Total Cholesterol, LDL-C, HDL-C, Triglycerides) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in fasting lipid profile to assess cardiometabolic effects of tirzepatide. All components of the lipid panel are measured in millimole/liter.
Liver Function Markers (Alanine transaminase, Alkaline phosphatase) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in liver enzymes to monitor hepatic safety. Hepatic enzymes are measured in Units per Litre.
Liver Function Markers (Bilirubin) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Changes in bilirubin to monitor hepatic safety. Bilirubin (Total, Direct, Indirect) are measured in micromoles per litre.
Cardiac Biomarkers (NT-proBNP) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Serum biomarker used to assess cardiac strain, providing insights into the broader metabolic effects of tirzepatide. NT-proBNP is measured in picograms per millilitre.
Inflammatory Biomarkers (hs-CRP) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Serum biomarkers used to assess inflammation providing insights into the broader metabolic effects of tirzepatide. hs-CRP is measured in milligrams per litre.
Inflammatory Biomarkers (IL-6) | At enrollment, Week 16, and Week 32, At Week 8 and Week 16 post-study.
  Serum biomarkers used to assess inflammation, providing insights into the broader metabolic effects of tirzepatide. IL-6 is measured in picograms per millilitre.
C-Peptide | At enrollment and at Week 32, At Week 8 and Week 16 post-study.
  Change in fasting C-peptide to assess residual β-cell function.
Carotid-Femoral Pulse Wave Velocity and Pulse Wave Analysis | At enrollment and at Week 32 (site-dependent).
  Measures of arterial stiffness and central blood pressure, used to evaluate vascular effects of treatment.
DXA Body Composition | At enrollment and at Week 32 (site-dependent).
  Whole-body DXA assessment of fat mass, lean mass, visceral fat, and bone density.
Echocardiogram (Diastolic Function Parameters) | At enrollment and at Week 32 (site-dependent).
  Assessment of cardiac structure and diastolic function, including E/A ratio, e', E/e', and left atrial volume.
VO₂-max Test | At enrollment and at Week 32 (site-dependent).
  Measurement of maximal oxygen consumption to evaluate cardiopulmonary fitness.
Quality-of-Life Measures (Diabetes Distress Scale) | At enrollment and at Week 32.
  Changes in the standardized Diabetes Distress Scale using the validated questionnaire. A participant's score is measured as the sum of responses to the appropriate items divided by the number of items in that scale.
  A mean item score 2.0 - 2.9 is considered moderate distress, and a mean item score > 3.0 is considered high distress.
Quality-of-Life Measures (Hypoglycemia Fear Survey II) | At enrollment and at Week 32.
  Changes in the standardized Hypoglycemia Fear Survey II using the validated questionnaire.
  HFS-II Total Score range: 0-132.
  Higher scores on the total HFS-II indicate a greater fear of hypoglycemia. The questionnaire does not have pre-defined cut-off scores for diagnostic categories; instead, the scores are used to measure the level of fear.
Quality-of-Life Measures (Three Factor Eating r18 Questionnaire) | At enrollment and at Week 32.
  Changes in the standardized Three Factor Eating Questionnaire scores.
  The three-factor eating questionnaire provides a score from 0 to 100 for cognitive restraint, uncontrolled eating, and emotional eating. Higher scores indicate greater cognitive restraint, uncontrolled eating, and emotional eating.
Gastric Emptying via [13C] Acetate Breath Test | At enrollment (or training visit) and at Week 32 (site-dependent).
  Rate of gastric emptying assessed by breath ¹³CO₂ appearance following standardized test meal.
Blood Glucagon Response to Standardized Meal | At enrollment and at Week 32 (site-dependent).
  Change in glucagon concentrations following ingestion of a standardized liquid meal.
Meal Tracking Using Keenoa or MyFood24 | Prior to randomization, during Week 16, and during Week 32.
  Assessment of caloric intake and macronutrient composition via 3-day dietary records.

OTHER OUTCOMES:
Severe hypoglycemia | From the time the participant signs informed consent until the end of study participation at Week 32, with additional safety follow-up at Week 8 and Week 16 post-study.
  Episode requiring the assistance of another person, due to altered consciousness, to administer carbohydrates, glucagon, or other resuscitative actions.
Diabetic Ketoacidosis | From the time the participant signs informed consent until the end of study participation at Week 32, with additional safety follow-up at Week 8 and Week 16 post-study.
  Clinical episode characterized by hyperglycemia/euglycemia, ketonemia or ketonuria, metabolic acidosis, and associated symptoms such as nausea, vomiting, abdominal pain, rapid breathing, or altered consciousness. Events requiring emergency evaluation, intravenous fluids, or hospital treatment will be recorded as DKA. All episodes will be assessed for severity, timing, precipitating factors, and their relationship to study interventions, including tirzepatide use and automated insulin delivery performance.
Gastrointestinal and related side effects | From the time the participant signs informed consent until the end of study participation at Week 32, with additional safety follow-up at Week 8 and Week 16 post-study.
  Nausea Vomiting Abdominal pain Diarrhea Constipation Liver profile changes Gallbladder disease Acute pancreatitis Other related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Melissa-Rosina Pasqua, MD-PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Ahmad Haidar, PhD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (2):
  - Institut de Recherches Cliniques de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Insel Hospital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data may be shared with qualified researchers after completion of the trial and publication of the primary results. Shared data may include de-identified demographic variables, glucose and insulin delivery data, laboratory results, questionnaire scores, and device-based assessments collected during the study. All data will be reviewed to minimize re-identification risk in accordance with Canadian and Swiss privacy regulations. Researchers must submit a scientifically valid proposal and sign a data use agreement. Requests will be reviewed by the study team, and approved data will be provided through a secure transfer process.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available beginning 12 months after publication of the primary results and for a period of five years thereafter.
Access Criteria: Researchers must submit a scientifically valid proposal and sign a data use agreement.

REFERENCES:
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Karlsson J, Persson LO, Sjostrom L, Sullivan M. Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. Int J Obes Relat Metab Disord. 2000 Dec;24(12):1715-25. doi: 10.1038/sj.ijo.0801442. PMID 11126230
- [Background] Saisho Y. Use of Diabetes Treatment Satisfaction Questionnaire in Diabetes Care: Importance of Patient-Reported Outcomes. Int J Environ Res Public Health. 2018 May 9;15(5):947. doi: 10.3390/ijerph15050947. PMID 29747423
- [Background] Gonder-Frederick LA, Schmidt KM, Vajda KA, Greear ML, Singh H, Shepard JA, Cox DJ. Psychometric properties of the hypoglycemia fear survey-ii for adults with type 1 diabetes. Diabetes Care. 2011 Apr;34(4):801-6. doi: 10.2337/dc10-1343. Epub 2011 Feb 23. PMID 21346182
- [Background] Fisher L, Hessler D, Polonsky W, Strycker L, Masharani U, Peters A. Diabetes distress in adults with type 1 diabetes: Prevalence, incidence and change over time. J Diabetes Complications. 2016 Aug;30(6):1123-8. doi: 10.1016/j.jdiacomp.2016.03.032. Epub 2016 Apr 4. PMID 27118163
- [Background] Frias JP, Davies MJ, Rosenstock J, Perez Manghi FC, Fernandez Lando L, Bergman BK, Liu B, Cui X, Brown K; SURPASS-2 Investigators. Tirzepatide versus Semaglutide Once Weekly in Patients with Type 2 Diabetes. N Engl J Med. 2021 Aug 5;385(6):503-515. doi: 10.1056/NEJMoa2107519. Epub 2021 Jun 25. PMID 34170647
- [Background] Martin C, Ravussin E, Sanchez-Delgado G, Nishiyama H, Li J, Urva S, et al. The effect of tirzepatide during weight loss on food intake, appetite, food preference and food craving in people with obesity. Can J Diabetes. 2023 Jul;47(7 Suppl):S199. doi:10.1016/j.jcjd.2023.10.370
- [Background] Snell-Bergeon JK, Kaur G, Renner D, Akturk HK, Beatson C, Garg SK. Effectiveness of Semaglutide and Tirzepatide in Overweight and Obese Adults with Type 1 Diabetes. Diabetes Technol Ther. 2025 Jan;27(1):1-9. doi: 10.1089/dia.2024.0328. Epub 2025 Jan 2. PMID 39745353
- [Background] Pasqua MR, Tsoukas MA, Kobayati A, Aboznadah W, Jafar A, Haidar A. Subcutaneous weekly semaglutide with automated insulin delivery in type 1 diabetes: a double-blind, randomized, crossover trial. Nat Med. 2025 Apr;31(4):1239-1245. doi: 10.1038/s41591-024-03463-z. Epub 2025 Jan 10. PMID 39794615
- [Background] Ahmann AJ, Capehorn M, Charpentier G, Dotta F, Henkel E, Lingvay I, Holst AG, Annett MP, Aroda VR. Efficacy and Safety of Once-Weekly Semaglutide Versus Exenatide ER in Subjects With Type 2 Diabetes (SUSTAIN 3): A 56-Week, Open-Label, Randomized Clinical Trial. Diabetes Care. 2018 Feb;41(2):258-266. doi: 10.2337/dc17-0417. Epub 2017 Dec 15. PMID 29246950
- [Background] Capehorn MS, Catarig AM, Furberg JK, Janez A, Price HC, Tadayon S, Verges B, Marre M. Efficacy and safety of once-weekly semaglutide 1.0mg vs once-daily liraglutide 1.2mg as add-on to 1-3 oral antidiabetic drugs in subjects with type 2 diabetes (SUSTAIN 10). Diabetes Metab. 2020 Apr;46(2):100-109. doi: 10.1016/j.diabet.2019.101117. Epub 2019 Sep 17. PMID 31539622
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Tsoukas MA, Cohen E, Legault L, von Oettingen JE, Yale JF, Vallis M, Odabassian M, El Fathi A, Rutkowski J, Jafar A, Ghanbari M, Gouchie-Provencher N, Rene J, Palisaitis E, Haidar A. Alleviating carbohydrate counting with a FiASP-plus-pramlintide closed-loop delivery system (artificial pancreas): Feasibility and pilot studies. Diabetes Obes Metab. 2021 Sep;23(9):2090-2098. doi: 10.1111/dom.14447. Epub 2021 Jun 21. PMID 34047449
- [Background] Karakus KE, Klein MP, Akturk HK, Shah VN. Changes in Basal and Bolus Insulin Requirements with Tirzepatide as an Adjunctive Therapy in Adults with Type 1 Diabetes Using Tandem Control-IQ. Diabetes Ther. 2024 Jul;15(7):1647-1655. doi: 10.1007/s13300-024-01592-9. Epub 2024 May 14. PMID 38743306
- [Background] Rivera Gutierrez R, Tama E, Bechenati D, Castaneda Hernandez R, Bennett PK, McNally AW, Fansa S, Anazco D, Acosta A, Hurtado Andrade MD. Effect of Tirzepatide on Body Weight and Diabetes Control in Adults With Type 1 Diabetes and Overweight or Obesity. Mayo Clin Proc. 2025 Feb;100(2):265-275. doi: 10.1016/j.mayocp.2024.07.006. Epub 2024 Nov 26. PMID 39601745
- [Background] Templer S. Closed-Loop Insulin Delivery Systems: Past, Present, and Future Directions. Front Endocrinol (Lausanne). 2022 Jun 6;13:919942. doi: 10.3389/fendo.2022.919942. eCollection 2022. PMID 35733769
- [Background] Meade LT, Rushton WE. Accuracy of Carbohydrate Counting in Adults. Clin Diabetes. 2016 Jul;34(3):142-7. doi: 10.2337/diaclin.34.3.142. PMID 27621531
- [Background] Weinzimer SA, Steil GM, Swan KL, Dziura J, Kurtz N, Tamborlane WV. Fully automated closed-loop insulin delivery versus semiautomated hybrid control in pediatric patients with type 1 diabetes using an artificial pancreas. Diabetes Care. 2008 May;31(5):934-9. doi: 10.2337/dc07-1967. Epub 2008 Feb 5. PMID 18252903
- [Background] Peacock S, Frizelle I, Hussain S. A Systematic Review of Commercial Hybrid Closed-Loop Automated Insulin Delivery Systems. Diabetes Ther. 2023 May;14(5):839-855. doi: 10.1007/s13300-023-01394-5. Epub 2023 Apr 5. PMID 37017916
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] Janez A, Guja C, Mitrakou A, Lalic N, Tankova T, Czupryniak L, Tabak AG, Prazny M, Martinka E, Smircic-Duvnjak L. Insulin Therapy in Adults with Type 1 Diabetes Mellitus: a Narrative Review. Diabetes Ther. 2020 Feb;11(2):387-409. doi: 10.1007/s13300-019-00743-7. Epub 2020 Jan 4. PMID 31902063
- See also: Mounjaro Monograph — https://pi.lilly.com/ca/mounjaro-ca-pmi.pdf